CLINICAL TRIAL: NCT03463629
Title: Multidisciplinary Team Approach: Working Together to Improve Glycemic Control in Hispanic Adults With Uncontrolled Type 2 Diabetes
Brief Title: Multidisciplinary Team Approach: Working Together to Improve Glycemic Control in Hispanic Adults Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: DHR Health Institute for Research and Development (Other)
Responsible Party: Principal Investigator, Mayra Judith Cantu, Family Nurse Practitioner, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SN-18-0075
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes
Keywords: Multidisciplinary Team; Hispanic adults
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specialized multidisciplinary diabetes team (SMDT) approach (Experimental): The implementation of the pilot study will consist of a specialized multidisciplinary diabetes team care (SMDT) that includes endocrinologists, a nurse practitioner, dieticians, pharmacists and a licensed professional counselors (LPCs) to collaborate and coordinate care. Subjects in the pilot study will follow a multidisciplinary team approach process with the following team members: pharmacist, LPC, and dietician.
  There will be 3 individualized visits: 1 visit with the counselor (LPC), 1 visit with the Pharmacist, and 1 visit with the Dietician.
  In addition, a follow up phone call post visit, that can range from 5 to 30 minutes, will be scheduled from each of the team members during the study. Also, throughout the pilot study participant's blood glucose readings will be monitored weekly via a transmittable wireless patient transmission monitor.
  Interventions: Other: Specialized multidisciplinary diabetes team (SMDT) approach
- Traditional model of care (Active Comparator): Receive the traditional model of care, but will not receive diabetes education by pharmacists or counseling services. Data for this arm will be collected through retrospective chart review.
  Interventions: Other: Traditional model of care

INTERVENTIONS:
Other: Specialized multidisciplinary diabetes team (SMDT) approach — The implementation of the pilot study will consist of a specialized multidisciplinary diabetes team care (SMDT) that includes endocrinologists, a nurse practitioner, dieticians, pharmacists and a licensed professional counselors (LPCs) to collaborate and coordinate care. Subjects in the pilot study will follow a multidisciplinary team approach process with the following team members: pharmacist, LPC, and dietician.
  There will be 3 individualized visits: 1 visit with the counselor (LPC), 1 visit with the Pharmacist, and 1 visit with the Dietician.
  In addition, a follow up phone call post visit, that can range from 5 to 30 minutes, will be scheduled from each of the team members during the study. Also, throughout the pilot study participant's blood glucose readings will be monitored weekly via a transmittable wireless patient transmission monitor.
  Arms: Specialized multidisciplinary diabetes team (SMDT) approach
Other: Traditional model of care — Receive the traditional model of care, but will not receive diabetes education by pharmacists or counseling services
  Arms: Traditional model of care

SUMMARY:
This study seeks to determine if a specialized multidisciplinary diabetes team (SMDT) approach that incorporates the use of the chronic care model can be an effective method for improving glycemic control in Hispanic adults with uncontrolled type 2 diabetes residing in the Rio Grande Valley. The study will expand the current model of care used and focus on the multidimensional aspects that consist of physical, nutritional, educational and psychological needs of this underserved Hispanic population residing in the Rio Grande Valley.

ELIGIBILITY:
Inclusion Criteria:

* Have physician-diagnosed type 2 diabetes
* Be self-identified as Hispanic or Latino
* An A1c value between 9-14% within the last three months
* English or Spanish speaking

Exclusion Criteria:

* Type 1 diabetes or gestational diabetes
* Cognitive impairment
* Prisoners or individuals under detention
* Unable to speak or understand English or Spanish
* Medical history of the end-stage renal disease or undergoing dialysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Change in glucose level as indicated by HbA1c levels | baseline, 3 months
  In this outcome, only the specialized multidisciplinary diabetes team (SMDT) arm (and not the traditional model of care arm) will be assessed.

SECONDARY OUTCOMES:
Change in patient satisfaction with a multidisciplinary team approach management as indicated by a diabetes treatment satisfaction questionnaire (DTSQ) | baseline, 3 months
Level of diabetes problem areas as assessed by the Problem Areas in Diabetes Questionnaire (PAID) questionnaire | baseline, 3 months
Change in body mass index (BMI) | baseline, 3 months
Change in weight | baseline, 3 months
Change in blood pressure | baseline, 3 months

OTHER OUTCOMES:
Glucose level as indicated by HbA1c levels | 3 months
  The objective of this outcome is to compare and evaluate HbA1c results from participants that received care through a multidisciplinary diabetes team with patients that have received only the traditional model of care.

CONTACTS AND LOCATIONS:
Overall Officials: Mayra J Cantu, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States